CLINICAL TRIAL: NCT04100733
Title: Surveillance of High-grade Non-muscle Invasive Bladder Tumours Using the Xpert Bladder Cancer Monitor
Acronym: SEALS Xpert
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jørgen Bjerggaard Jensen (Other)
Collaborators: Cepheid (Industry)
Responsible Party: Sponsor-Investigator, Jørgen Bjerggaard Jensen, Professor, consultant, Aarhus University Hospital
Organization: Aarhus University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SEALS Xpert
Record Dates: First submitted 2019-09-19; First posted 2019-09-24 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Non-muscle Invasive Bladder Cancer; Urinary Biomarker
Keywords: Flexible cystoscopy; Xpert Bladder Cancer Monitor
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Study subjects will cohere to current clinical guidelines for follow-up regimes of HG NMIBC with flexible cystoscopy and cytology every four months for a period of two years.
  Interventions: Diagnostic Test: Flexible cystoscopy (WL/NBI) and urinary cytology
- Intervention (Experimental): Patients in the interventional arm will be followed at 4, 8, 16 and 20 months after inclusion with Xpert Bladder Cancer Monitor-test (and urinary cytology) instead of flexible cystoscopy.
  Interventions: Diagnostic Test: Xpert Bladder Cancer Monitor

INTERVENTIONS:
Diagnostic Test: Xpert Bladder Cancer Monitor — Xpert Bladder Cancer Monitor detects mRNA fragments from 5 genes frequently overexpressed in non-muscle invasive bladder cancer.
  Arms: Intervention
Diagnostic Test: Flexible cystoscopy (WL/NBI) and urinary cytology — Adhering to current danish guidelines for follow-up of non-muscle invasive bladder cancer.
  Arms: Control

SUMMARY:
The study aims to evaluate the potential clinical impact of a highly sensitive urinary marker, the Xpert Bladder Cancer Monitor, regarding possible reduction in number of flexible cystoscopies in an outpatient setting without decreasing recurrence-free survival or increasing risk of progression.

DETAILED DESCRIPTION:
Epidemiology and treatment Bladder cancer is the 12th most diagnosed cancer worldwide with an incidence of approximately 550 000 new cases each year.1 A majority of the tumors are characterized as non-muscle invasive bladder cancer (NMIBC), meaning stage T1 according to the 2016 TNM-classification.2 Treatment of primary NMIBC is transurethral resection of the bladder (TUR-B) and treatment of recurring NMIBC is repeated TUR-B and often adjuvant instillation therapy with either Mitomycin C or Bacillus Calmette-Geerin (BCG) according to the histology of the tumor. NMIBC-tumors are graded into high grade (HG) and low grade (LG) according to the histological characteristics of their TUR-B specimen. Generally, intravesical Mitomycin C is recommended to treat LG tumors and intravesical BCG is recommended for treating HG tumors.3,4.

Follow-up schedules based on risk of recurrence. The histological grade, number of tumors, tumor size, T-stage, recurrence-rate and presence of carcinoma in situ (CIS) is used to estimate risk of recurrence according to the EORTC-scoring system. Based on the risk stratification, different follow-up schedules after initial TUR-B are planned. High risk tumors are followed-up with flexible cystoscopy and urinary cytology every four months until two recurrence-free years, whereas low and intermediate risk tumors are followed utilizing the 4-8-12 model where intervals between follow up are increased for patients without recurrence until 5 disease-free years.3 The evidence behind these follow-up schedules is not based on high level evidence and research but rather on tradition and 'clinical experience'.

Clinical challenge of current follow-up schedules The majority of patients with HG tumors will have recurrence despite treatment, especially within the two first years after diagnosis. Moreover, many patients will receive lifelong follow-up cystoscopy and urinary cytology tests. Follow-up schedules are costly due to many visits at the hospital for flexible cystoscopy, urinary cytology, and treatment. A micro-costing analysis performed by the Urological Research Unit at Aarhus University Hospital prior to initiation of the current study, has shown that the total expense in relation to flexible cystoscopy in the outpatient clinic is approximately 315 EUR per examination (Appendix 1). Equally important to frequency and cost of follow-up, every follow-up visit is associated with patient discomfort, pain, risk of infections, and strictures of the urethra.6 Each cystoscopy carries a 15% risk of complications. Nearly 1,500 cystoscopies are carried out in HG patients in Central Denmark Region each year, resulting in approximately 240 complications each year, with cystitis being the most common complication. Furthermore, flexible cystoscopy is not always reliable in terms of diagnosing recurrences and CIS.7-9

Urinary biomarkers A proposed alternative to flexible cystoscopy in the detection of recurrent NMBIC is non-invasive molecular urinary markers that detect mRNA, protein or DNA from selected genes relevant for bladder cancer in urine samples. Several studies have been prospectively validated and shown high sensitivity and specificity for urinary markers.10,11 Recently, the Xpert Bladder Cancer Monitor test was shown by Valenberg et al.12 to have a sensitivity of 83% and specificity of 76% for HG disease and similarly D'Elia et al.13 showed a specificity of 77% and sensitivity of 46% for a cohort of mainly LG patients. However, studies have until now focused mainly on detection of NMIBC in patients with incident tumors, which are most often larger and more easily diagnosed with urinary biomarkers than recurrences.14 To our knowledge, no studies have so far substituted cystoscopies for urinary biomarkers in a randomized controlled setting. Thus, the need for high level evidence regarding the use of urinary biomarkers for surveillance of NMIBC is still there.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years of age at the time of signing the Informed Consent Form
* Ability to understand the Participant Information sheet orally and in writing
* Signed Informed Consent Form
* Is, according to the investigator's judgement, able to comply with the trial protocol
* Previously diagnosed with high grade NMIBC Recurrence free at the time of inclusion detected by flexible cystoscopy

Exclusion Criteria:

* History of any upper urinary tract tumor regardless of grade and stage within the last 5 years prior to randomization
* T1 tumor where re-resection has not been performed
* CIS or invasive tumor within 3 months before randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 392 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Recurrence-free survival | 2 years follow-up per patient
  Time from inclusion to detection of recurrence of bladder cancer.

CONTACTS AND LOCATIONS:
Locations (3):
- Denmark (3):
  - Hospital of West Jutland, Holstebro, Danmark
  - Aarhus University Hospital, Århus N
  - Zealand University Hospital, Roskilde